CLINICAL TRIAL: NCT06382064
Title: Evaluation of Wear Experience With PRECISION7® Contact Lenses in Habitual Acuvue® Oasys® Lens Wearers
Brief Title: Evaluation of Wear Experience With One Week Reusable Contact Lenses in Habitual Two Week Reusable Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Fogt, Principal Investigator, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024H0089
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Myopia
Keywords: Contact Lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Subjects will be fit into Acuvue Oasys contact lenses at the first visit to wear for 2 weeks. Subjects will then be fit into PRECISION7 lenses at the second visit to wear for 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contact Lens Wear Experience (Experimental): Participants will be enrolled in the study for 4 weeks. Biweekly replacement contact lenses will be worn for the first 2 weeks. One-week replacement lenses worn for second 2 weeks.
  Interventions: Device: Biweekly replacement contact lenses; Device: One week replacement contact lenses

INTERVENTIONS:
Device: Biweekly replacement contact lenses — Biweekly replacement reusable contact lenses.
Device: One week replacement contact lenses — One week replacement reusable contact lenses.

SUMMARY:
This open-label study is of current Acuvue® Oasys® wearers (2 - week replacement, reusable lenses) who are satisfied with their current lenses. Subjects will be refit into one week reusable contact lenses and will wear lenses for approximately 2 weeks. Subjects will return for vision and lens fit assessments and will complete surveys about their wear experience.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Ability to give informed consent
3. Current Acuvue® Oasys® spherical lens wearer.
4. Distance visual acuity of 20/25 or better with current contact lenses in each eye.
5. Good general health defined by, medication use that has not changed within the last 30 days and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the Investigator.
6. Willing to spend time for the study, which includes: attend three study visits and wear contact lenses on days between study visits.

Exclusion Criteria:

1. Current or active ocular inflammation or infection as determined by the Investigator.
2. Currently pregnant or lactating. (Participants will be asked to self-report these conditions).
3. Systemic inflammatory disease (i.e. Diabetes, etc.) that could confound study results in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contact Lens Wear Experience
Started | 71
Completed | 62
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Contact Lens Wear Experience
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 44
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjective Assessment of Lens Wear Experience
Description: Subjective assessment of lens wear experience using a CLDEQ-8 survey (contact lens dry eye questionnaire). There are 8 questions about about the presence and intensity of symptoms when wearing contact lenses. When totaling the scores for each question, the lowest possible score=1 and the highest possible score=37. Higher scores result from more prevalent and intense symptoms.
Time Frame: After 2 weeks of wear in the 1-week replacement reusable lenses.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Contact Lens Wear Experience
Number analyzed (Participants) | 62
Scores on a scale | 10 [6 to 16]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Contact Lens Wear Experience
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT06382064/Prot_SAP_001.pdf